CLINICAL TRIAL: NCT03294954
Title: GD2 Specific Chimeric Antigen Receptor (CAR) and Interleukin-15 Expressing Autologous Natural Killer T-cells to Treat Children With Neuroblastoma
Brief Title: GD2 Specific CAR and Interleukin-15 Expressing Autologous NKT Cells to Treat Children With Neuroblastoma
Acronym: GINAKIT2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Gengwen Tian, MD, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-41033 GINAKIT2
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Natural Killer T-Cells; Chimerical Antigen Receptor
MeSH Terms: conditions — Neuroblastoma | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GINAKIT cells (Experimental): GINAKIT cells will be administer to patients with Neuroblastomas on Day 0.
  Interventions: Genetic: GINAKIT Cells
- Experimental: GINAKIT cells + Etanercept. (Experimental): GINAKIT cells will be administer to patients with Neuroblastomas on Day 0 in combination of Etanercept.
  Interventions: Biological: GINAKIT cells + Etanercept

INTERVENTIONS:
Genetic: GINAKIT Cells — Six dose levels of GINAKIT cells will be studied. Dosing will be based on the actual number of transduced cells. All doses are per m2.
  * Dose Level 1 = 3 x 10^6
  * Dose Level 2 = 1 x 10^7
  * Dose Level 3 = 3 x 10^7
  * Dose Level 4 = 1 x 10^8
  * Dose Level 5 = 3 x 10^8
  * Dose Level 6 = 1 x 10^9
  Arms: GINAKIT cells
Biological: GINAKIT cells + Etanercept — Four dose levels of GINAKIT cells in combination of Etanercept will be studied. Dosing will be based on the actual number of transduced cells. All doses are per m2.
  * Combination Dose level 1: 3 x 10^6 + Etanercept*
  * Combination Dose level 2: 1 x 10^7 + Etanercept*
  * Combination Dose level 3: 3 x 10^7 + Etanercept*
  * Combination Dose level 4: 1 x 10^8 + Etanercept
  Arms: Experimental: GINAKIT cells + Etanercept.

SUMMARY:
This research study combines two different ways of fighting cancer: antibodies and Natural Killer T cells (NKT). Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special white blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. Investigators have found from previous research that they can put a new gene into T cells that will make them recognize cancer cells and kill them. In a previous clinical trial, investigators made artificial genes called a chimeric antigen receptors (CAR), from an antibody called 14g2a that recognizes GD2, a molecule found on almost all neuroblastoma cells (GD2-CAR). Investigators put these genes into the patients' own T cells and gave them back to patients that had neuroblastoma.

NKT cells are another special subgroup of white blood cells that can specifically go into tumor tissue of neuroblastoma. Inside the tumor, there are other white blood cells called macrophages which help the cancer cells to grow and recover from injury. NKT cells can specifically kill these macrophages and slow the tumor growth.

We will expand NKT cells and add GD2-specific chimeric antigen receptors to the cells. We think these cells might be better able to attack NB since they also work by destroying the macrophages that allows the tumor to grow. The chimeric antigen receptor will also contain a gene segment to make the NKT cells last longer. This gene segment is called CD28. In addition, to further improve the antitumor activity of the GINAKIT cells we added another gene expressing a molecule called Interleukin -15 (IL-15). The combination of these 3 components showed the most antitumor activity by CAR expressing NKT cells and improved these cells' survival in animal models. We also found that a medicine called ETANercept can slow down neuroblastoma growth, which might enhance the effects of the modified cells. In this part of our study, we aim to treat children with hard-to-treat neuroblastoma using these modified NKT cells along with ETANercept. Though ETANercept has been used to treat other diseases, such as rheumatoid arthritis in children, there is limited information about the safety, efficacy, and risk of ETANercept treatment in combination with cellular therapies.

GD2-CAR expressing NKTs have not been tested in patients so far. The purpose of this study is to find the largest effective and safe dose of GD2-CAR NKT cells (GINAKIT cells), to evaluate their effect on the tumor and how long they can be detected in the patient's blood and what affect they have on the patient's neuroblastoma.

DETAILED DESCRIPTION:
In this study the first step is to collect blood from the patient to make the GINAKIT cells. Once the GINAKIT cells are made they will be administered to the patient.

Patients will be treated on a single fixed dose level with Etanercept from now on. If there is severe toxicity related to the combination of GINAKIT cells and Etanercept, we will treat patients on lower dose level. Thus maximum 36 patients will be recruited on the on the combination therapy, including 18 patients potentially at the lower dose level. If we are not able to generate sufficient GINAKIT cells on the fixed dose level, we will treat you with the highest dose level that is achieved.

Before getting the GINAKIT cells, the patient will receive cyclophosphamide and fludarabine intravenously (through a needle inserted into a vein or a port-a-cath) for 2 days and then fludarabine alone for one more day. The patient will then receive ETANercept subcutaneously (through a needle just under the skin) once per week starting the day after chemotherapy for 5 doses. The patient will receive the GINAKIT cells the day after first dose of ETANercept.

The patient will be given an injection of GINAKIT cells into the vein through an IV line at the assigned dose. Before the patient receives the injection, they may be given a dose of Benadryl (diphenhydramine) and Tylenol (acetaminophen). The injection will take up to 10 minutes. The patient will be monitored in the clinic after the injection for about 4 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital.

The patient will need to stay in Houston for 4 weeks after the infusion so investigators can monitor the patient for side effects. The patient will have follow-up visits (at weeks 1, 2, 3, 4 and 8; months 3, 6, 9, and 12; twice a year for 4 years and then once a year for the next 10 years - for a total of 15 years) and scheduled disease evaluations after the GINAKIT cell infusion (at week 6 and then as clinically needed).

If after 4 weeks the patient's condition does not get worse, the patient may receive another round of lymphodepleting chemotherapy and infusion of GINAKIT2 cells. Reinfusion of cells may occur up to three times and the patient will have to meet treatment eligibility criteria at each lymphodepletion start. The patient will also receive ETANercept with the schedule at each time of treatment. Treatment eligibility are characteristics that must be met such as current health status and other items that ensure patients who could be made worse by participating in the study are not exposed to that risk. The eligibility also ensures researchers achieve accurate results

Before being treated, the patient will receive a series of standard medical tests as follows:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function
* Blood tests to ensure the patient do not have tuberculosis.
* Buccal swabs (cheek scraping)
* Measurements of the patient's tumor by routine imaging studies and bone marrow evaluation within 4 weeks (preferably 2 weeks) before start of lymphodepletion (no other cancer treatment should be given after these studies and the GINAKIT cell infusion). Imaging studies that have been used in the past to best assess the patient's tumor will be used (Computer Tomogram (CT) or Magnetic Resonance Imaging (MRI), and Positron Emission Tomography (PET/CT), and/or MIBG scan). A PET scan is an imaging test that uses radioactive material to look for disease in the body. A MIBG scan is an imaging test that uses radioactive material and a special scanner to find or confirm the presence of neuroblastoma.
* A urine pregnancy test. If that patient is pregnant both the patient and their parents will be informed of the pregnancy.

The patient will receive standard medical tests when they are getting the infusions and afterwards as follows:

* Physical exams
* Blood tests to measure blood cells counts, kidney and liver function.
* Subcutaneous injection of ETANercept.
* Measurements of the patient's tumor by routine imaging studies 4-6 weeks after the infusion.
* Tumor biopsy at 2 weeks and between 4-6 weeks after the infusion and as clinically indicated thereafter. The evaluation at week 2 after the infusion is for research only and is done to see whether or not there are GINAKIT cells in the tumor. For all clinically indicated tumor biopsies a portion of the sample for research will be requested.
* If a tumor was in the bone marrow at the time of treatment, the procedure will be repeated at 2 weeks and between 4-6 weeks after the infusion and as clinically indicated thereafter. The evaluation at week 2 after the infusion is for research only and is done to see whether or not there are GINAKIT cells in the bone marrow. For all clinically indicated bone marrow collections a portion of the sample for research will be requested.

To learn more about the way the GINAKIT cells are working and how long they last in the body, an extra amount of blood will be obtained before the chemotherapy, on the day of the GINAKIT cell infusion (before and at the end of the infusion), 1, 2, 3, 4 and 8 weeks after the GINAKIT cell infusion, every 3 months for the 1st year, every 6 months for the next 4 years and then once a year for the next 10 years (for a total of 15 years). The amount of blood taken will be based on the patient's weight with up to a maximum of 60 ml (12 teaspoons) of blood to be obtained at any one time. For children, the total amount of blood drawn will not be more than 3 ml (less than 1 teaspoon) per 1 kg of body weight on any given day. This volume is considered safe, but may be decreased if the patient is anemic (have a low red blood cell count). This blood will also be used to monitor the patient's white blood cell levels. In the event the patient's white blood cell counts are high, they will be admitted to the hospital where they will be treated with hydration, steroids or chemotherapy. The study doctor will discuss with the patient the best treatment options.

During the time points listed above, if the GINAKIT cells are found in the patient's blood at a certain amount, an extra 5ml of blood may need to be collected for additional testing.

If the patient has a procedure where tumor samples are obtained, investigators will request a sample to be used for research purposes.

If the patient develops a second abnormal growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested (if a sample can be obtained).

The patient will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

Because the patient will receive cells with a new gene in them they will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

ELIGIBILITY:
Procurement Inclusion Criteria:

1. Relapsed or refractory high risk neuroblastoma
2. Life expectancy of at least 12 weeks
3. Age greater than 1 year and less than 21 years old
4. Karnofsky/Lansky score of 60% or greater
5. Absence of HAMA prior to enrollment (only in patients that have been previously treated with murine antibodies)
6. Ability to tolerate leukocyte apheresis
7. Informed consent and assent (as applicable) obtained from parent/guardian and child.
8. Patients must have an ANC greater than or equal to 500/µl, platelet count greater than or equal to 20,000/µl. Patients may be transfused to obtain a platelet count greater than or equal to 20,000/µl.
9. Pulse Ox greater than or equal to 90% on room air
10. Serum AST less than 3 times the upper limit of normal
11. Total Bilirubin less than 1.5 times the upper limit of normal
12. Creatinine < 1.5 times the upper limit of normal
13. Recovered from the acute toxic effects of all prior chemotherapy based on the enrolling physician's assessment (if some effects of chemotherapy are expected to last long term, patient is eligible if meeting other eligibility criteria).
14. Weight greater than 12kg
15. Negative QuantiFERON-TB or T-SPOT testing within 3 months prior to procurement

Procurement Exclusion Criteria:

1. Rapidly progressive disease
2. History or hypersensitivity to murine protein-containing products
3. Tumor causing airway obstruction
4. Currently receiving immunosuppressive drugs such as corticosteroids, tacrolimus or cyclosporine
5. Severe previous toxicity from cyclophosphamide or fludarabine based on the enrolling physician's assessment
6. HIV infection
7. History of hypersensitivity, anaphylaxis, and/or adverse event with Etanercept

Treatment Inclusion Criteria:

1. Relapsed or refractory high risk neuroblastoma
2. Life expectancy of at least 12 weeks
3. Age greater than 1 year and less than 21 years old
4. Karnofsky/Lansky score of 60% or greater
5. Patients must have an ANC greater than or equal to 500/µl, platelet count greater than or equal to 20,000/µl. Patients may be transfused to obtain a platelet count greater than or equal to 20,000/µl.
6. Pulse Ox greater than or equal to 90% on room air
7. Serum AST less than 3 times the upper limit of normal
8. Total Bilirubin less than 1.5 times the upper limit of normal
9. Creatinine < 1.5 times the upper limit of normal
10. Recovered from the acute toxic effects of all prior chemotherapy based on the enrolling physician's assessment (if some effects of chemotherapy are expected to last long term, patient is eligible if meeting other eligibility criteria and expected to tolerate lymphodepletion).
11. Absence of human anti-mouse antibodies (HAMA) prior to enrollment for patients who have received prior therapy with murine antibodies
12. Patients must have autologous transduced NKTs with greater than or equal to 20% expression of GD2-specific CAR.
13. Informed consent and assent (as applicable) obtained from parent/guardian and child.
14. Weight greater than 12kg
15. Negative QuantiFERON-TB or T-SPOT testing within 3 months prior to the start of LD

Treatment Exclusion Criteria:

1. Rapidly progressive disease
2. Currently receiving any investigational drugs
3. History or hypersensitivity to murine protein-containing products
4. Cardiomegaly or bilateral pulmonary infiltrates on chest radiograph or CT. However, patients with cardiomegaly on imaging may be enrolled if they have an assessment of cardiac function (i.e., ECHO or MUGA) within 3 weeks of starting protocol therapy that is within normal limits. Additionally, patients with bilateral pulmonary infiltrates on imaging may be enrolled if the lesions are not consistent with active neuroblastoma (i.e., negative on functional imaging with PET or MIBG, or by pathologic assessment).
5. Tumor potentially causing airway obstruction
6. Pregnancy or lactation or not willing to use birth control
7. Currently receiving immunosuppressive drugs such as corticosteroids, tacrolimus or cyclosporine
8. Severe previous toxicity form cyclophosphamide or fludarabine based on the enrolling physician's assessment
9. HIV infection
10. History of hypersensitivity, anaphylaxis, and/or adverse event with Etanercept

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2040-08-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of autologous NKTs expressing a 2nd generation GD2-specific chimeric antigen receptor administered to patients with relapsed or refractory neuroblastoma in combination with Etanercept. | 28 days
  Defined as the highest dose level that will have at most a 33% chance of inducing the following NKT-cell-related dose limiting toxicities (DLTs) within 28 days after infusion of NKTs in combination with Etanercept.

SECONDARY OUTCOMES:
Anti-tumor response of autologous GINAKIT cells in patients with relapsed/refractory neuroblastoma and compare the anti-tumor response in patients treated with and without Etanercept. | 15 years
  Summarize tumor response by calculating overall response rates and report the Kaplan-Meier curves for the relapse-free survival.

OTHER OUTCOMES:
Immunologic response of autologous GINAKIT cells with and without Etanercept in patients with relapsed/refractory neuroblastoma. | 15 years
  Summarize at pre- and post-infusion time points using descriptive statistics to evaluate their expansion and persistence. Changes in each of these NKTs in combination with Etanercept from pre-infusion to each time point of post-infusion will be assessed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Gengwen Tian, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Heczey A, Xu X, Courtney AN, Tian G, Barragan GA, Guo L, Amador CM, Ghatwai N, Rathi P, Wood MS, Li Y, Zhang C, Demberg T, Di Pierro EJ, Sher AC, Zhang H, Mehta B, Thakkar SG, Grilley B, Wang T, Weiss BD, Montalbano A, Subramaniam M, Xu C, Sachar C, Wells DK, Dotti G, Metelitsa LS. Anti-GD2 CAR-NKT cells in relapsed or refractory neuroblastoma: updated phase 1 trial interim results. Nat Med. 2023 Jun;29(6):1379-1388. doi: 10.1038/s41591-023-02363-y. Epub 2023 May 15. PMID 37188782
- [Derived] Heczey A, Courtney AN, Montalbano A, Robinson S, Liu K, Li M, Ghatwai N, Dakhova O, Liu B, Raveh-Sadka T, Chauvin-Fleurence CN, Xu X, Ngai H, Di Pierro EJ, Savoldo B, Dotti G, Metelitsa LS. Anti-GD2 CAR-NKT cells in patients with relapsed or refractory neuroblastoma: an interim analysis. Nat Med. 2020 Nov;26(11):1686-1690. doi: 10.1038/s41591-020-1074-2. Epub 2020 Oct 12. PMID 33046868
- [Derived] Xu X, Huang W, Heczey A, Liu D, Guo L, Wood M, Jin J, Courtney AN, Liu B, Di Pierro EJ, Hicks J, Barragan GA, Ngai H, Chen Y, Savoldo B, Dotti G, Metelitsa LS. NKT Cells Coexpressing a GD2-Specific Chimeric Antigen Receptor and IL15 Show Enhanced In Vivo Persistence and Antitumor Activity against Neuroblastoma. Clin Cancer Res. 2019 Dec 1;25(23):7126-7138. doi: 10.1158/1078-0432.CCR-19-0421. Epub 2019 Sep 4. PMID 31484667